CLINICAL TRIAL: NCT00884494
Title: Role of Ghrelin in the Improvement of Insulin Resistance After Roux-en-Y Gastric Bypass Surgery
Brief Title: Ghrelin and Insulin Resistance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Robyn Tamboli, Research Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB#090362; NIH: RO1-DK070860-01S1
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Insulin Resistance; Normal Weight,Healthy Controls
Keywords: Obesity; Insulin resistance; Ghrelin
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y gastric bypass (Experimental)
  Interventions: Drug: Ghrelin infusion to assess effects on insulin sensitivity
- Lean (Experimental)
  Interventions: Drug: Ghrelin infusion to assess effects on insulin sensitivity

INTERVENTIONS:
Drug: Ghrelin infusion to assess effects on insulin sensitivity

SUMMARY:
Ghrelin, a hormone produced in the stomach that stimulates hunger and food intake, declines immediately after weight loss surgery. Some studies suggest that ghrelin may worsen an individual's ability to respond to insulin. The purpose of this study is to determine if the decline in ghrelin levels after weight loss surgery contributes to the improvement of insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria for RYGB group:

* Age 18-65
* BMI > 35 kg/m2
* Scheduled for bariatric surgery at Vanderbilt University Medical Center

Inclusion Criteria for Lean group:

* Age 18-65
* BMI < 30kg/m2

Exclusion Criteria:

* Prior bariatric surgery
* Serum creatinine > 1.5 mg/dl
* Hepatic enzyme elevations > 2x upper limits of normal
* Current use of warfarin or clopidogrel
* Intercurrent infections
* Females with positive pregnancy test
* Abnormal ECG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of ghrelin on insulin resistance in obese subject, as well as subjects in the immediate post-RYGB period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Tamboli, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji Abumrad, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Garcia AE, Kasim N, Tamboli RA, Gonzalez RS, Antoun J, Eckert EA, Marks-Shulman PA, Dunn J, Wattacheril J, Wallen T, Abumrad NN, Flynn CR. Lipoprotein Profiles in Class III Obese Caucasian and African American Women with Nonalcoholic Fatty Liver Disease. PLoS One. 2015 Nov 23;10(11):e0142676. doi: 10.1371/journal.pone.0142676. eCollection 2015. PMID 26599819